CLINICAL TRIAL: NCT00810056
Title: Fostering Healthy Futures Efficacy Trial for Preadolescent Youth in Foster Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Kempe Foundation for the Prevention and Treatment of Child Abuse and Neglect (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 02-0516b; R01MH076919 (NIH)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Child Abuse
Keywords: Child abuse and neglect; Out-of-home care; Mentoring; Skills groups; Assessment
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assessment only (Active Comparator): Cognitive, academic achievement and mental health screening assessment and report.
  Interventions: Other: Assessment
- Assessment + FHF (Experimental): Cognitive, academic achievement and mental health screening assessment and report. Fostering Healthy Futures program (FHF) including weekly therapeutic skill groups and mentoring over a 9-month period.
  Interventions: Other: Assessment; Behavioral: Fostering Healthy Futures (FHF)

INTERVENTIONS:
Other: Assessment — Cognitive, academic achievement, and mental health screening assessment and report.
Behavioral: Fostering Healthy Futures (FHF) — Weekly therapeutic skill groups and mentoring over a 9-month period.
  Arms: Assessment + FHF

SUMMARY:
This is a multi-county randomized controlled trial of the Fostering Healthy Futures (FHF) preventive intervention program (consisting of mentoring and skills groups) with 256 maltreated preadolescent youth in out-of-home care. It is hypothesized that participation in the FHF program will result in better functioning in cognitive, social, and behavioral domains, and that these gains will result in improved mental health functioning, quality of life, and reductions in problem behaviors and adverse life-course outcomes.

DETAILED DESCRIPTION:
Youth with a history of maltreatment and foster care placement are at risk for a host of mental health, behavioral, and social problems, resulting in adverse life-course outcomes of great public health significance. This is a 5-year efficacy trial of the Fostering Healthy Futures Program (FHF), a preventive intervention designed to promote prosocial development, and to reduce problem behaviors for youth in foster care. FHF is an innovative, culturally-sensitive and multi-component intervention for 9-11-year-old children who have been maltreated and placed in foster care. Through a 9-month intervention that includes screening assessments, one-on-one mentoring, and skills groups, FHF targets cognitive, social and behavioral domains in order to build competencies, improve mental health functioning and quality of life, and reduce problem behaviors and adverse life outcomes (e.g. arrests, school dropout, restrictive placements). Assessments with youth, caregivers and teachers will be conducted at baseline (pre-randomization), post-intervention, and 1-year follow-up. Data will also include child welfare, educational, and juvenile justice records. A randomized controlled pilot trial of FHF in one county has produced program manuals for the mentoring and skills group components, and evidence of program feasibility, with high recruitment and retention rates. The FHF pilot study has demonstrated positive preliminary effects on putative mediators. A multi-county randomized controlled trial of the FHF program with 256 youth will enable the investigators to: 1) examine intervention effects on both proximal and distal outcomes, 2) examine potential moderators of the intervention, 3) conduct mediational analyses to identify the mechanisms by which the program may enhance outcomes, and 4) conduct within-group analyses. The goal is to design more efficacious interventions, thereby reducing disability, morbidity, and mortality, not only for youth in foster care, but for all high-risk youth.

ELIGIBILITY:
Inclusion Criteria:

All of the 9-11-year-old children court-ordered into out-of-home care (as a result of maltreatment) over the prior year in participating counties, including:

1. Youth placed in group homes, foster homes, and with kin
2. Youth with significant behavior problems
3. Youth who meet criteria for mental health diagnoses or dual diagnosis
4. Youth with mild cognitive impairment

Exclusion Criteria:

1. Youth who reunify before the beginning of the intervention
2. Youth with significant cognitive, behavioral, and/or mental health impairment that interfered with either with their ability to benefit from the prevention program or to participate safely
3. Youth who were not proficient enough in English to participate
4. Youth who lived too far (more than 35 minutes) from sites where groups were held

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 426 (Actual)
Dates: Start 2007-06; Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of Child mental health, social, & behavioral functioning and quality of life as measured from multiple informants and sources. | 6 and 16 months post intervention

SECONDARY OUTCOMES:
Evaluation of Problem behaviors, life-course outcomes, placement history, and service system involvement as measured from multiple informants and sources. | 6 and 16 months post intervention and possible future timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Heather N Taussig, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver, Adams, Arapahoe, Jeferson and Broomfield Counties, Denver, Colorado, United States

REFERENCES:
- [Background] Taussig HN, Culhane SE, Hettleman D. Fostering healthy futures: an innovative preventive intervention for preadolescent youth in out-of-home care. Child Welfare. 2007 Sep-Oct;86(5):113-31. PMID 18422051
- [Derived] Hambrick E, Lee SK, Weiler L, Collins JO, Rhodes T, Taussig H. Engagement in a Preventive Intervention for Preadolescent Children in Foster Care: Considerations for Intervention Design. Child Psychiatry Hum Dev. 2023 Oct;54(5):1373-1385. doi: 10.1007/s10578-022-01341-8. Epub 2022 Mar 18. PMID 35303199
- [Derived] Taussig HN, Dmitrieva J, Garrido EF, Cooley JL, Crites E. Fostering Healthy Futures Preventive Intervention for Children in Foster Care: Long-term Delinquency Outcomes from a Randomized Controlled Trial. Prev Sci. 2021 Nov;22(8):1120-1133. doi: 10.1007/s11121-021-01235-6. Epub 2021 Apr 27. PMID 33905053